CLINICAL TRIAL: NCT03973996
Title: Gut-level Antiinflammatory Activities of Green Tea in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Bruno, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2018H0592
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Dysbiosis; Endotoxemia; Metabolic Syndrome; Inflammation
Keywords: Green tea; Gut barrier function; Gut dysbiosis; Inflammation; Metabolic endotoxemia; Metabolic syndrome; Microbiome
MeSH Terms: conditions — Dysbiosis; Endotoxemia; Metabolic Syndrome; Inflammation | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green Tea (Experimental): Participants consuming gummy confections with catechin-rich green tea extract daily for 4 weeks
  Interventions: Dietary Supplement: Green Tea Extract
- Placebo (Placebo Comparator): Participants consuming matched gummy confections formulated without green tea extract daily for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Green Tea Extract — A gummy confection with catechin-rich green tea extract (1 g/d)
  Other Names: Camellia sinesis plant extract
  Arms: Green Tea
Dietary Supplement: Placebo — A matched gummy confection formulated without green tea extract
  Arms: Placebo

SUMMARY:
This study evaluates dietary green tea extract to improve gut health and inflammation in persons with metabolic syndrome and healthy adults. Participants will complete two phases of intervention in random order in which they will consume green tea extract or placebo for one month and then switch to the opposite treatment for an additional month.

DETAILED DESCRIPTION:
Tea is the most abundantly consumed prepared beverage in the world. Green tea, containing catechins, exerts antiinflammatory activities. However, a fundamental gap exists concerning its intestinal-level targets that can prevent metabolic syndrome (MetS) development and progression. Studies in obese rodents indicate that green tea inhibits nuclear factor kappa-light-chain-enhancer of activated B cells (NFκB) activation by limiting gut-derived endotoxin translocation to the portal circulation and decreasing hepatic Toll-like receptor-4 (TLR4) pro-inflammatory signaling. The objective of this clinical investigation is to establish evidence-based recommendations for green tea, based on improvements in endotoxemia and restored gut barrier function, that promote optimal health. The hypothesis is that green tea catechins function to limit metabolic endotoxemia by ameliorating gut dysbiosis-mediated inflammation that otherwise provokes intestinal permeability. This will be tested by conducting a double-blind, placebo-controlled, randomized-order, crossover trial in MetS and healthy persons to examine the efficacy of green tea on metabolic endotoxemia. Each treatment will be one-month in duration and separated by a washout period. The anticipated outcomes are expected to be of significance, because they will advance a dietary strategy to help avert MetS complications attributed to metabolic endotoxemia by establishing antiinflammatory prebiotic and antimicrobial bioactivities of catechins that promote intestinal health.

ELIGIBILITY:
Inclusion criteria:

Individuals with ≥3 of the following established criteria for metabolic syndrome:

* Fasting glucose 100-126 mg/dL
* Waist circumference >89/>102 cm for females/males
* HDL-C <50/<40 mg/dL for females/males
* Triglyceride >150 mg/dL
* Blood pressure >130/85 mmHg

Healthy adults:

* Body weight 19-25 kg/m2
* Fasting glucose <100 mg/dL
* HDL-C >50/>40 mg/dL for females/males
* Triglyceride <150 mg/dL
* Blood pressure <120/80 mmHg

Exclusion criteria:

* Concurrent tea consumption
* Use of dietary supplements, prebiotics, or probiotics
* Use of antibiotics or antiinflammatory agents
* History of liver disease, cardiovascular disease, hypertension (blood pressure >140/90 mmHg), or cancer
* History of gastrointestinal disorders, chronic diarrhea, or surgeries
* Hemochromatosis
* Parkinson's disease
* Use of medications to manage diabetes, hypertension, or hyperlipidemia
* Use of antipsychotic medications [Clozapine, lithium, Diazepam]
* Use of blood thinning medications [Warfarin]
* Use of high blood pressure medications [nadolol]
* Use of monoamine oxidase inhibitors [selegiline]
* Alcohol consumption >2 drinks/d
* Smoking tobacco
* Vegetarian
* Pregnancy, lactation, or recent changes in birth control use for women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Bruno, PhD, RD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dey P, Sasaki GY, Wei P, Li J, Wang L, Zhu J, McTigue D, Yu Z, Bruno RS. Green tea extract prevents obesity in male mice by alleviating gut dysbiosis in association with improved intestinal barrier function that limits endotoxin translocation and adipose inflammation. J Nutr Biochem. 2019 May;67:78-89. doi: 10.1016/j.jnutbio.2019.01.017. Epub 2019 Feb 8. PMID 30856467
- [Background] Li J, Sasaki GY, Dey P, Chitchumroonchokchai C, Labyk AN, McDonald JD, Kim JB, Bruno RS. Green tea extract protects against hepatic NFkappaB activation along the gut-liver axis in diet-induced obese mice with nonalcoholic steatohepatitis by reducing endotoxin and TLR4/MyD88 signaling. J Nutr Biochem. 2018 Mar;53:58-65. doi: 10.1016/j.jnutbio.2017.10.016. Epub 2017 Nov 3. PMID 29190550
- [Background] Hodges JK, Zhu J, Yu Z, Vodovotz Y, Brock G, Sasaki GY, Dey P, Bruno RS. Intestinal-level anti-inflammatory bioactivities of catechin-rich green tea: Rationale, design, and methods of a double-blind, randomized, placebo-controlled crossover trial in metabolic syndrome and healthy adults. Contemp Clin Trials Commun. 2019 Nov 20;17:100495. doi: 10.1016/j.conctc.2019.100495. eCollection 2020 Mar. PMID 31799477
- [Result] Zeng M, Hodges JK, Pokala A, Khalafi M, Sasaki GY, Pierson J, Cao S, Brock G, Yu Z, Zhu J, Vodovotz Y, Bruno RS. A green tea extract confection decreases circulating endotoxin and fasting glucose by improving gut barrier function but without affecting systemic inflammation: A double-blind, placebo-controlled randomized trial in healthy adults and adults with metabolic syndrome. Nutr Res. 2024 Apr;124:94-110. doi: 10.1016/j.nutres.2024.02.001. Epub 2024 Feb 5. PMID 38430822

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy - Placebo Then GTE: Participants with normal metabolic health will consume placebo gummy confections (formulated without green tea extract) daily for 4 weeks, followed by a 4-week washout period, and then consume catechin-rich green tea extract (1 g/day) gummy confections daily for 4 weeks.
- MetS - GTE Then Placebo: Participants with metabolic syndrome will consume catechin-rich green tea extract (1 g/day) gummy confections daily for 4 weeks, followed by a 4-week washout period, and then consume placebo gummy confections (formulated without green tea extract) daily for 4 weeks.
- Healthy- GTE Then Placebo: Participants with normal metabolic health will consume catechin-rich green tea extract (1 g/day) gummy confections daily for 4 weeks, followed by a 4-week washout period, and then consume placebo gummy confections (formulated without green tea extract) daily for 4 weeks.
- MetS - Placebo Then GTE: Participants with metabolic syndrome will consume placebo gummy confections (formulated without green tea extract) daily for 4 weeks, followed by a 4-week washout period, and then consume catechin-rich green tea extract (1 g/day) gummy confections daily for 4 weeks.
Period: First Intervention (4 Weeks)
Arm/Group | Healthy - Placebo Then GTE | MetS - GTE Then Placebo | Healthy- GTE Then Placebo | MetS - Placebo Then GTE
Started | 10 | 12 | 11 | 13
Completed | 9 | 11 | 10 | 10
Not Completed | 1 | 1 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 3
Period: Washout (4 Weeks)
Arm/Group | Healthy - Placebo Then GTE | MetS - GTE Then Placebo | Healthy- GTE Then Placebo | MetS - Placebo Then GTE
Started | 9 | 11 | 10 | 10
Completed | 9 | 11 | 10 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Healthy - Placebo Then GTE | MetS - GTE Then Placebo | Healthy- GTE Then Placebo | MetS - Placebo Then GTE
Started | 9 | 11 | 10 | 10
Completed | 9 | 11 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy-Placebo Then GTE: Participants with normal metabolic health will consume placebo gummy confections (formulated without green tea extract) daily for 4 weeks, followed by a 4-week washout period, and then consume catechin-rich green tea extract (1 g/day) gummy confections daily for 4 weeks.
- MetS- Placebo Then GTE: Participants with metabolic syndrome will consume placebo gummy confections (formulated without green tea extract) daily for 4 weeks, followed by a 4-week washout period, and then consume catechin-rich green tea extract (1 g/day) gummy confections daily for 4 week
- MetS- GTE Then Placebo: Participants with metabolic syndrome will consume catechin-rich green tea extract (1 g/day) gummy confections daily for 4 weeks, followed by a 4-week washout period, and then consume placebo gummy confections (formulated without green tea extract) daily for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Healthy-Placebo Then GTE | Healthy- GTE Then Placebo | MetS- Placebo Then GTE | MetS- GTE Then Placebo | Total
Number analyzed (Participants) | 9 | 10 | 10 | 11 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 10 | 11 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 5 | 8 | 25
  Male | 4 | 3 | 5 | 3 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 10 | 11 | 40
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21.5 (1.3) | 23.1 (2.1) | 36.9 (5.5) | 33.7 (3.2) | 29.1 (7.4)
Fasting blood glucose [Mean (Standard Deviation); unit: mg/dL] | 87.1 (5.6) | 91.0 (5.9) | 105.0 (6.5) | 100.2 (10.3) | 96.1 (10.1)
Fasting triglycerides [Mean (Standard Deviation); unit: mg/dL] | 47.2 (16.8) | 73.5 (24.1) | 132.7 (66.1) | 199.5 (83.1) | 117.0 (81.0)
Fasting HDL [Mean (Standard Deviation); unit: mg/dL] | 64.3 (17.5) | 59.2 (12.7) | 42.3 (11.9) | 36.1 (5.6) | 49.7 (16.7)
Waist circumference [Mean (Standard Deviation); unit: cm] | 77.4 (4.3) | 79.1 (6.9) | 114.7 (10.9) | 109.6 (12.4) | 96.0 (19.4)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 115.4 (5.8) | 113.5 (7.6) | 125.5 (7.6) | 121.9 (10.4) | 119.3 (9.2)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 74.6 (3.5) | 74.7 (5.7) | 85.0 (8.1) | 83.8 (6.8) | 79.8 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Serum Endotoxin
Description: Data are biomarker fasting concentrations.
Time Frame: Day 28
Measure: Mean (Standard Error); unit: EU/mL
Groups:
- Healthy - Placebo; MetS - Placebo; MetS - GTE: Confection without green tea extract consumed daily for 4 weeks.
- Healthy - GTE: Confection with green tea extract consumed daily for 4 weeks.
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
EU/mL | 31.6 (2.5) | 26.7 (2.6) | 44.5 (2.4) | 39.1 (2.5)

2. Secondary Outcome: Plasma Lipopolysaccharide-binding Protein
Description: Data are biomarker fasting concentrations
Time Frame: Day 28
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
ng/mL | 4035 (339) | 4435 (380) | 7890 (1143) | 8572 (1394)

3. Secondary Outcome: Urinary Lactulose/Mannitol Ratio
Description: Lactulose/mannitol ratio in urine collected 0-5 h post-ingestion of non-digestible sugar probes.
Time Frame: Day 28
Measure: Mean (Standard Error); unit: ratio
Groups:
- Healthy - GTE; MetS - GTE: Participants consuming gummy confections with catechin-rich green tea extract daily for 4 weeks
  Green Tea Extract: A gummy confection with catechin-rich green tea extract (1 g/d)
- Healthy - Placebo; MetS - Placebo: Participants consuming matched gummy confections formulated without green tea extract daily for 4 weeks
  Placebo: A matched gummy confection formulated without green tea extract
Arm/Group | Healthy - GTE | Healthy - Placebo | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
ratio | 0.075 (0.009) | 0.084 (0.012) | 0.087 (0.013) | 0.065 (0.007)

4. Secondary Outcome: Urinary Sucralose/Erythritol Ratio
Description: Sucralose/Erythritol ratio measured in urine collected 0-24 h post-ingestion of non-digestible sugar probes
Time Frame: Day 28
Measure: Mean (Standard Error); unit: ratio
Groups:
- MetS - GTE: Confection with green tea extract consumed daily for 4 weeks.
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
ratio | 0.014 (0.0014) | 0.014 (0.0015) | 0.015 (0.001) | 0.015 (0.001)

5. Secondary Outcome: Plasma Interleukin-6
Description: Data are biomarker concentrations at fasting
Time Frame: Day 28
Measure: Mean (Standard Error); unit: pg/mL
Groups:
- Healthy - GTE; MetS - GTE: Participants consumed gummy confections with catechin-rich green tea extract daily for 4 weeks
  Green Tea Extract: A gummy confection with catechin-rich green tea extract (1 g/d)
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
pg/mL | 1.9 (0.085) | 1.9 (0.070) | 3.1 (0.24) | 3.3 (0.29)

6. Secondary Outcome: Fecal Calprotectin
Description: Data are biomarker fecal concentrations, measured in samples pooled from specimens collected on Days 25-27 of the 28-day intervention.
Time Frame: Day 25-27 (pooled samples) of the 28-day intervention
Measure: Mean (Standard Error); unit: ug/g
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
ug/g | 35.9 (5.5) | 24.4 (2.7) | 42.5 (9.3) | 36.7 (5.2)

7. Secondary Outcome: Fecal Myeloperoxidase
Description: as for outcome 6
Time Frame: Day 25-27 (pooled samples) of the 28-day intervention
Measure: Mean (Standard Error); unit: ng/g
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
ng/g | 97.4 (9.9) | 83.4 (7.5) | 148.1 (40.9) | 97.9 (10.5)

8. Secondary Outcome: Plasma Epigallocatechin Gallate
Description: Data are plasma concentrations of epigallocatechin gallate
Time Frame: Day 28
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/L | 0.001 (0.001) | 0.343 (0.057) | 0.00 (0.00) | 0.21 (0.04)

9. Secondary Outcome: Plasma Epicatechin
Description: Data are plasma concentrations of epicatechin.
Time Frame: Day 28
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/L | 0.0 (0.0) | 0.022 (0.0048) | 0.00016 (0.00016) | 0.015 (0.003)

10. Secondary Outcome: Plasma Epicatechin Gallate
Description: Data are plasma concentrations of epicatechin gallate.
Time Frame: Day 28
Measure: Mean (Standard Error); unit: umol/L
Groups:
- Healthy - GTE; MetS - GTE: Participants consumed gummy confections with catechin-rich green tea extract daily for 4 weeks.
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/L | 0.002 (0.001) | 0.30 (0.037) | 0.002 (0.001) | 0.20 (0.027)

11. Secondary Outcome: Plasma 3,4-γ-valerolactone
Description: Data are biomarker concentrations at fasting
Time Frame: Day 28
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/L | 0.008 (0.005) | 0.17 (0.050) | 0.007 (0.003) | 0.090 (0.031)

12. Secondary Outcome: Plasma 3,4,5-γ-Valerolactone
Description: Data are biomarker concentrations at fasting
Time Frame: Day 28
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/L | 0.001 (0.001) | 0.034 (0.017) | 0.0017 (0.0010) | 0.0060 (0.0047)

13. Secondary Outcome: Plasma Soluble Cluster of Differentiation-14
Description: Data are biomarker concentrations at fasting
Time Frame: Day 28
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
ng/mL | 1465 (57) | 1459 (71) | 1424 (67) | 1367 (83)

14. Secondary Outcome: Plasma Glucose
Description: Data are biomarker concentrations at fasting
Time Frame: Day 28
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
mg/dL | 86.3 (1.6) | 83.9 (1.5) | 98.9 (3.0) | 98.6 (2.6)

15. Secondary Outcome: Plasma Insulin
Description: Data are biomarker concentrations at fasting
Time Frame: Day 28
Measure: Mean (Standard Error); unit: μIU/mL
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
μIU/mL | 6.4 (0.7) | 6.0 (0.6) | 19.6 (2.3) | 22.4 (3.8)

16. Secondary Outcome: Plasma Triglyceride
Description: Data are biomarker concentrations at fasting
Time Frame: Day 28
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
mg/dL | 51.2 (4.1) | 54.7 (4.9) | 140.5 (14.0) | 149.9 (17.0)

17. Secondary Outcome: Plasma Total Cholesterol
Description: Data are biomarker concentrations at fasting
Time Frame: Day 28
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
mg/dL | 195.5 (9.4) | 186.9 (6.7) | 220.1 (9.0) | 215.6 (10.2)

18. Secondary Outcome: Serum Alanine Transaminase
Description: Data are biomarker concentrations at fasting
Time Frame: Day 28
Measure: Mean (Standard Error); unit: (U/L)
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
(U/L) | 15.0 (0.9) | 15.0 (1.0) | 24.2 (2.1) | 23.6 (2.3)

19. Secondary Outcome: Serum Aspartate Transaminase
Description: Data are biomarker concentrations at fasting
Time Frame: Day 28
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
U/L | 17.3 (0.9) | 17.5 (0.8) | 19.5 (0.8) | 20.2 (1.0)

20. Secondary Outcome: Blood Hematocrit
Description: Data are biomarker concentrations at fasting
Time Frame: Day 28
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
Percent | 44.3 (0.7) | 45.1 (0.8) | 44.0 (0.6) | 43.5 (0.6)

21. Secondary Outcome: Plasma Tumor Necrosis Factor-alpha
Description: Data are biomarker fasting concentrations
Time Frame: Day 28
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
pg/mL | 1.2 (0.32) | 2.3 (0.53) | 4.8 (0.81) | 5.0 (0.62)

22. Secondary Outcome: Fecal Butyrate
Description: Data are biomarker concentrations in fecal samples, measured in samples pooled from specimens collected on Days 25-27 of the 28-day intervention.
Time Frame: Days 25-27 (pooled samples) of the 28-day intervention
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/g | 11.7 (1.8) | 10.8 (1.4) | 16.6 (2.4) | 13.9 (1.4)

23. Secondary Outcome: Fecal Acetate
Description: as for outcome 22
Time Frame: Days 25-27 (pooled samples) of the 28-day intervention
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/g | 35.9 (5.2) | 33.1 (3.4) | 47.9 (4.1) | 41.9 (3.5)

24. Secondary Outcome: Fecal Valeric Acid
Description: as for outcome 22
Time Frame: Day 25-27 (pooled samples) from the 28-day intervention
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/g | 0.95 (0.16) | 0.91 (0.13) | 2.04 (0.30) | 1.86 (0.25)

25. Secondary Outcome: Fecal Hexanoic Acid
Description: as for outcome 22
Time Frame: Day 25-27 (pooled samples) from the 28-day intervention
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/g | 0.56 (0.16) | 0.49 (0.14) | 0.98 (0.59) | 0.55 (0.32)

26. Secondary Outcome: Fecal Isobutyric Acid
Description: as for outcome 22
Time Frame: Day 25-27 (pooled samples) from the 28-day intervention
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/g | 1.86 (0.18) | 1.67 (0.22) | 1.87 (0.21) | 1.87 (0.15)

27. Secondary Outcome: Fecal 2-Methylbutyric
Description: as for outcome 22
Time Frame: Day 25-27 (pooled samples) of the 28-day intervention
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/g | 1.29 (0.13) | 1.14 (0.16) | 1.20 (0.15) | 1.20 (0.11)

28. Secondary Outcome: Fecal Isovaleric Acid
Description: as for outcome 22
Time Frame: Day 25-27 (pooled samples) of the 28-day intervention
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/g | 1.40 (0.14) | 1.22 (0.16) | 1.38 (0.16) | 1.40 (0.12)

29. Secondary Outcome: Plasma Ascorbic Acid
Description: Data are biomarker fasting concentrations
Time Frame: Day 28
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/L | 40.2 (4.7) | 41.6 (4.3) | 32.1 (4.5) | 28.6 (3.6)

30. Secondary Outcome: Plasma Uric Acid
Description: Data are biomarker fasting concentrations
Time Frame: Day 28
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Healthy - Placebo | Healthy - GTE | MetS - Placebo | MetS - GTE
Number analyzed (Participants) | 19 | 19 | 21 | 21
umol/L | 244.7 (13.8) | 256.0 (14.0) | 330.3 (13.9) | 319.8 (16.0)

ADVERSE EVENTS:
Time Frame: One month for each intervention
Description: Includes all participants who received at least one dose of intervention
Groups:
- Healthy Participants - GTE Confection Intervention; MetS Participants - GTE Confection Intervention: Participants received GTE confections 3-times daily for 1-month, instructed to take with meals
- Healthy Participants - Placebo Confection Intervention; MetS Participants - Placebo Confection Intervention: Participants received Placebo confections 3-times daily for 1-month, instructed to take with meals
Arm/Group | Healthy Participants - GTE Confection Intervention | Healthy Participants - Placebo Confection Intervention | MetS Participants - GTE Confection Intervention | MetS Participants - Placebo Confection Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/22 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT03973996/Prot_SAP_000.pdf